CLINICAL TRIAL: NCT00002133
Title: An Open Study of the Effect of Itraconazole Oral Solution for the Treatment of Fluconazole Refractory Oropharyngeal Candidiasis in HIV-Positive Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janssen, LP (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 236B; ITR-USA-94
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: Itraconazole; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Candidiasis, Oral
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Itraconazole

INTERVENTIONS:
Drug: Itraconazole

SUMMARY:
To assess the efficacy and safety of itraconazole oral solution in HIV-seropositive patients with oropharyngeal candidiasis that is refractory to fluconazole.

DETAILED DESCRIPTION:
Patients receive itraconazole oral solution twice daily. Per 08/15/94 amendment, patients with complete resolution of oropharyngeal candidiasis lesions upon completion of treatment are eligible for maintenance treatment on protocol FDA 236C. Patients who decline maintenance are followed for 6 weeks. Patients who relapse during follow-up are re-treated for 14-28 days; if lesions clear, patients may enter the maintenance protocol.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV antibody seropositivity or diagnosis of AIDS.
* Confirmed oropharyngeal candidiasis.
* Failed fluconazole treatment within the past 14 days.
* Life expectancy of at least 3 months.
* NO symptoms of esophageal candidiasis (e.g., dysphagia) unless endoscopic exam of esophagus was performed and fungal esophagitis was not present.
* NO prior disseminated candidiasis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Underlying clinical condition that precludes study completion or places the patient at significant risk.
* Considered unreliable about following physician's directives.

Concurrent Medication:

Excluded:

* Investigational drugs (approved expanded access drugs are permitted).
* Rifampin.
* Rifabutin.
* Phenobarbital.
* Phenytoin.
* Carbamazepine.
* Terfenadine.
* Astemizole.

Patients with the following prior conditions are excluded:

* History of hypersensitivity to imidazole or azole compounds.
* Clinical evidence of significant hepatic disease within the past 2 months.

Prior Medication:

Excluded:

* Investigational drugs within 1 month prior to study entry (approved expanded access drugs are permitted).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Arkansas for Med Sciences, Little Rock, Arkansas
  - East Bay AIDS Ctr, Berkeley, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - Dr Douglas Ward, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - Infectious Diseases Research Clinic / Indiana Univ Hosp, Indianapolis, Indiana
  - Natl Inst of Allergy & Infect Dis / Cln Ctr, Bethesda, Maryland
  - Ann Arbor Veterans Administration Med Ctr, Ann Arbor, Michigan
  - Wayne State Univ / Harper Hosp, Detroit, Michigan
  - Washington Univ, St Louis, Missouri
  - Ohio State Univ Hosp, Columbus, Ohio
  - Oklahoma City Veterans Administration Med Ctr, Oklahoma City, Oklahoma
  - Pennsylvania Hosp, Philadelphia, Pennsylvania
  - Infectious Disease Clinic, Nashville, Tennessee
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas
  - Univ of Virginia Health Sciences Ctr, Charlottesville, Virginia

REFERENCES:
- [Background] Moskovitz B, Wu J, Baruch A, Benken C. Long term safety and efficacy of itraconazole oral solution (IS) for treatment of fluconazole refractory oropharyngeal candidiasis (OC) in HIV-positive patients (pts). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:124 (abstract no 325)